CLINICAL TRIAL: NCT01995188
Title: A Phase Ib, Open-Label, Dose-Escalation Study of the Safety and Pharmacology of DNIB0600A in Combination With Carboplatin (With or Without Bevacizumab) in Patients With Platinum-Sensitive Ovarian Cancer or Non-Squamous Non-small Cell Lung Cancer
Brief Title: A Study to Evaluate the Safety and Pharmacology of DNIB0600A in Participants With Platinum-Sensitive Ovarian Cancer or Non-Squamous Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GO29006
Record Dates: First submitted 2013-11-15; First posted 2013-11-26 (Estimated); Last update posted 2017-10-04 (Actual); Status verified 2017-10

CONDITIONS: Non-Squamous Non-Small Cell Lung Cancer
MeSH Terms: interventions — Bevacizumab; Carboplatin; lifastuzumab vedotin

ARMS (4):
- Dose Escalation Cohort: DNIB0600A+Carboplatin (Experimental): DNIB0600A at an initial dose of 1.2 milligrams per kilogram (mg/kg) will be administered via intravenous (IV) infusion further following a dose-escalation until DLT under consultation of the investigator in combination with Carboplatin fixed dose of area under the curve (AUC)=6 mg/milliliter(mL)*minute (min) administered by IV infusion on Day 1 of a 21-day cycle.
  Interventions: Drug: Carboplatin; Drug: DNIB0600A
- NSCLC Dose Expansion Cohort: DNIB0600A+Carboplatin (Experimental): Recommended phase 2 dose (RP2D) of DNIB0600A administered via IV infusion in combination with Carboplatin, AUC=6 mg/mL*min administered via IV infusion on Day 1 of each 21-day cycle in participants with NSCLC until disease progression or death, whichever occurs first.
  Interventions: Drug: DNIB0600A
- PSOC Dose Expansion Cohort: DNIB0600A+Carboplatin (Experimental): RP2D of DNIB0600A administered via IV infusion in combination with AUC=6 mg/mL*min administered via IV infusion on Day 1 of each 21-day cycle in participants with PSOC until disease progression or death, whichever occurs first.
  Interventions: Drug: Carboplatin; Drug: DNIB0600A
- PSOC Dose Expansion Cohort: DNIB0600A+Carboplatin+Bevacizumab (Experimental): RP2D of DNIB0600A administered via IV infusion in combination with Carboplatin, AUC=6 mg/mL*min and Bevacizumab 15 milligrams per kilogram (mg/kg) administered via IV infusion on Day 1 of each 21-day cycle in participants with PSOC until disease progression or death, whichever occurs first.
  Interventions: Drug: Bevacizumab; Drug: Carboplatin; Drug: DNIB0600A

INTERVENTIONS:
Drug: Bevacizumab — Bevacizumab 15 milligrams per kilogram (mg/kg) administered via IV infusion on Day 1 of each 21-day cycle until disease progression or death, whichever occurs first.
  Other Names: Avastin
  Arms: PSOC Dose Expansion Cohort: DNIB0600A+Carboplatin+Bevacizumab
Drug: Carboplatin — Carboplatin fixed dose of AUC=6 mg/mL*min administered by IV infusion on Day 1 of each 21-day dose escalation and expansion cycles. Carboplatin will be administered for a maximum of 6 cycles or until disease progression or unacceptable toxicity, whichever is first.
  Arms: Dose Escalation Cohort: DNIB0600A+Carboplatin; PSOC Dose Expansion Cohort: DNIB0600A+Carboplatin; PSOC Dose Expansion Cohort: DNIB0600A+Carboplatin+Bevacizumab
Drug: DNIB0600A — DNIB0600A at an initial dose of 1.2 mg/kg will be administered via IV infusion further following a dose-escalation until DLT under consultation of the investigator on Day 1 of 21 day dose-escalation cycle. RP2D will be administered further in dose-expansion for until disease progression or death, whichever occurs first.

SUMMARY:
This open-label, multicenter, phase 1b study will evaluate the safety and pharmacokinetics of DNIB0600A in participants with platinum-sensitive ovarian cancer (PSOC) or Non-Squamous Non-small Cell Lung Cancer (NSCLC). The maximum tolerated dose of intravenously infused DNIB0600A in combination with carboplatin will be determined in escalating dose cohorts. The combination of DNIB0600A and carboplatin will then be evaluated with and without bevacizumab [Avastin] in three dose expansion cohorts.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) status of 0 or 1.
* Histologically documented epithelial ovarian cancer, primary peritoneal cancer, or fallopian tube cancer that is platinum sensitive.
* PSOC (i.e., epithelial ovarian cancer, primary peritoneal cancer, or fallopian tube cancer) with documented radiographic progression or relapse within 6 to 18 months of most recent platinum-based chemotherapy.
* Female participants of childbearing potential must use effective contraception as defined by study protocol and cannot be pregnant or breastfeeding.

NSCLC-specific Inclusion Criteria:

* Histological documentation of incurable, locally advanced, or metastatic non-squamous
* NSCLC that has progressed on prior treatment
* Not more than 2 prior regimens in the metastatic setting, including one prior cytotoxic regimen and one prior non-cytotoxic regimen (prior treatment with adjuvant therapy within 6 months of recurrence is considered a treatment regimen in the metastatic setting).
* For participants with a documented epidermal growth factor receptor (EGFR) mutation or anaplastic lymphoma kinase (ALK) rearrangement, one additional line of non-cytotoxic prior treatment will be permitted provided the therapy is a targeted agent against the EGFR mutation or ALK rearrangement.
* For participants with lung cancer, centrally confirmed high expression of a sodium-dependent phosphate transporter (NaPi2b) by immunohistochemistry (IHC) is required (i.e., IHC 2+ or 3+).

Exclusion Criteria:

* Anti-tumor therapy of any kind or major surgery within 4 weeks prior to Day 1.
* For ovarian cancer participants only, platinum-based chemotherapy within 6 months prior to Day 1.
* For ovarian cancer participants only, platinum treatment with more than two platinum-based chemotherapy regiments or more than four anti-cancer regimens, overall, for the treatment of ovarian cancer.
* Palliative radiation within 2 weeks prior to Day 1.
* Toxicity (except alopecia and anorexia) from prior therapy or neuropathy of grades > 1.
* Evidence of any significant disease or condition that could affect compliance with the protocol or interpretation of results.
* Known active infection (except fungal nail infections).
* History of liver disease or human immunodeficiency virus (HIV).
* Other malignancy within the last 5 years, except for adequately treated or controlled carcinoma in situ of the cervix or skin cancer or primary endometrial cancer of stage </= 1B.
* Untreated or active central nervous system (CNS) metastases.
* Prior treatment with NaPi2b- targeted therapy.

Bevacizumab-Specific Exclusion Criteria (for Participants in Second Ovarian

Expansion Cohort Only):

* Inadequately controlled hypertension or history of hypertensive crisis or encephalopathy.
* History of heart problems or thrombosis within 6 months prior to study start.
* History of stroke within 6 months prior to study enrollment.
* History of significant vascular disease.
* History of expectoration of blood within 1 month prior to study start or blood clotting problems.
* Core biopsy or other minor surgical procedure within 7 days prior to study start
* Serious and non-healing wound, active ulcer, or untreated bone fracture.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2013-12-16 (Actual); Primary Completion 2016-11-09 (Actual); Study Completion 2016-11-09 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Dose-limiting Toxicities (DLTs) | 21 days
Number of Participants with Adverse events (AE) and Serious Adverse Events (SAEs) | Day 1 until 30 days after the last-infusion (up to approximately 3 years)
Number of Participants with Anti-DNIB0600A Antibodies | Pre-infusion (0 hour) at Day 1 of Cycle 1, 2, 3, 4 (each cycle of 21 days), 30 days after last infusion (up to approximately 3 years)

SECONDARY OUTCOMES:
Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - inf)] of DNIB0600A | Pre-infusion (0 hour), hour 0.5,1 post-infusion Cycle 1 (each cycle= 28 days); 7, 14 days post-infusion of Cycle 1 (Day 8, 15 respectively); Day 1 of Cycle 2 and subsequent cycles up to last dose; 30 days after last dose (up to approximately 3 years)
Maximum Observed Plasma Concentration (Cmax) | Pre-infusion (0 hour), hour 0.5,1 post-infusion Cycle 1 (each cycle= 28 days); 7, 14 days post-infusion of Cycle 1 (Day 8, 15 respectively); Day 1 of Cycle 2 and subsequent cycles up to last dose; 30 days after last dose (up to approximately 3 years)
Minimum Observed Plasma Trough Concentration (Cmin) | Pre-infusion (0 hour), hour 0.5,1 post-infusion Cycle 1 (each cycle= 28 days); 7, 14 days post-infusion of Cycle 1 (Day 8, 15 respectively); Day 1 of Cycle 2 and subsequent cycles up to last dose; 30 days after last dose (up to approximately 3 years)
Systemic Clearance (CL) | Pre-infusion (0 hour), hour 0.5,1 post-infusion Cycle 1 (each cycle= 28 days); 7, 14 days post-infusion of Cycle 1 (Day 8, 15 respectively); Day 1 of Cycle 2 and subsequent cycles up to last dose; 30 days after last dose (up to approximately 3 years)
Volume of Distribution at Steady State (Vss) | Pre-infusion (0 hour), hour 0.5,1 post-infusion Cycle 1 (each cycle= 28 days); 7, 14 days post-infusion of Cycle 1 (Day 8, 15 respectively); Day 1 of Cycle 2 and subsequent cycles up to last dose; 30 days after last dose (up to approximately 3 years)
Plasma Decay Half-Life (t1/2) | Pre-infusion (0 hour), hour 0.5,1 post-infusion Cycle 1 (each cycle= 28 days); 7, 14 days post-infusion of Cycle 1 (Day 8, 15 respectively); Day 1 of Cycle 2 and subsequent cycles up to last dose; 30 days after last dose (up to approximately 3 years)
Percentage of Participants With Objective Response as Assessed by Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) | From screening thereafter every 2 cycles (from Cycle 2 to Cycle 16) or every 4 cycles (from Cycle 10) until disease progression or death (up to approximately 3 years)
Duration of Objective Response Rate as Assessed by RECIST v1.1 | From screening thereafter every 2 cycles (from Cycle 2 to Cycle 16) or every 4 cycles (from Cycle 10) until disease progression or death (up to approximately 3 years)
Progression Free Survival (PFS) as Assessed by RECIST v1.1 | Day 1 to the first occurrence of disease progression or death within 30 days of the last administration of study drug, whichever occurs first (up to approximately 3 years)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (4):
- United States (4):
  - Massachusetts General Hospital., Boston, Massachusetts
  - Dana Farber Cancer Inst., Boston, Massachusetts
  - The University of Oklahoma, Oklahoma City, Oklahoma
  - The Sarah Cannon Research Inst, Nashville, Tennessee